CLINICAL TRIAL: NCT04852692
Title: A Retrospective/Prospective, Multicenter, Non-interventional, Historical Control Study Investigating Comparative Effectiveness of IMBRUVICA in Steroid Dependent/Refractory cGVHD Patients
Brief Title: A Study to Investigate the Comparative Effectiveness of Ibrutinib in Steroid Dependent/Refractory cGVHD Participants
Status: Terminated | Type: Observational
Why Stopped: After conducting pilot phase, the study team decided to stop the study as the study couldn't meet the study target number of patients and study objectives.
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108945; 54179060GVH4001 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Chronic Graft vs Host Disease
Keywords: Chronic; Ibrutinib; Retrospective; Prospective
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Part A: Retrospective Phase: Retrospective collection of data for eligible participants with steroid dependent/refractory chronic graft versus host disease (cGVHD) who initiated salvage treatments from initiation point (administration starting point of the salvage treatment) of the identified last-line of conventional salvage therapy for cGVHD treatment as their second-forth line therapy and will be collected for up to 24 weeks from the initiation point.
- Part B: Prospective Phase: Prospectively enroll participants with steroid dependent/refractory cGVHD that are decided to be treated with ibrutinib in second-fourth line therapy for the treatment of cGVHD. Participants will continue to receive corticosteroids as a standard of care.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of ibrutinib compared to conventional salvage treatments in participants with steroid dependent/refractory chronic graft versus host disease (cGVHD) by measuring overall cGVHD response (modified National Institutes of Health [NIH] response defined complete response [CR] and partial response [PR]) at Week 24.

ELIGIBILITY:
Inclusion Criteria:

Part A and Part B

* Must have a confirmed diagnosis of steroid dependent or refractory classic cGVHD defined at any time post-hematopoietic cell transplantation (HCT) as: a) refractory disease - progressive cGVHD manifestations requiring prednisolone at greater than or equal to (>=) 1 milligram per kilogram per day (mg/kg/day) for at least 1 week or persist without improvement despite continued treatment with glucocorticoid (prednisolone at >= 0.5 mg/kg/day or 1 mg/kg every other day) for at least 4 weeks; b) dependent disease: persistent cGVHD manifestations requiring glucocorticoid >= prednisolone 0.25 mg/kg/day or >=0.5mg/kg every other day for at least 8 weeks Part A
* Treated at least 2 or more therapies for cGVHD (including glucocorticoids)
* Participants whose identified last line of conventional salvage treatment is second-fourth line of therapy
* Index date (initiation date of the identified last-line of conventional salvage therapy) at least 28 weeks before the study initiation date Part B
* Treated at least 3 lines therapies for cGVHD (including glucocorticoids)
* Participants who are treated with ibrutinib in their second-fourth line of therapy

Exclusion Criteria:

Part A and Part B

* Known or suspected active acute GVHD
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 28 days Part A
* Treated with an investigational agent for their identified last-line of conventional salvage therapy
* Pregnant, breastfeeding during last-line of conventional salvage therapy Part B
* Pregnant, breast-feeding, or of childbearing potential without a negative serum or urine pregnancy test within 7 days of enrollment. Male or female participants of childbearing potential unwilling to use effective contraceptive precautions throughout the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with steroid dependent or refractory chronic graft versus host disease (cGVHD) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Percentage of Participants with Overall Response Rate | Week 24
  Overall response rate is defined as the percentage of participants who achieve complete response (CR) or partial response (PR) according to modified National Institutes of Health (NIH) response.

SECONDARY OUTCOMES:
Part B: Rate of Sustained Response | At least 5 months (up to 36 weeks)
  Sustained response rate will be assessed.
Part B: Duration of Response | Up to 5 months
  Duration of response will be assessed.
Part A and Part B: Corticosteroid Requirement Changes Over Time | Up to 24 weeks
  The change of the corticosteroid dose requirement during the treatment will be assessed.
Part B: Time to cGVHD Progression | Up to 36 weeks
  Time to chronic graft versus host disease (cGVHD) progression is defined as the time from the first dose of the ibrutinib to modified NIH response defined progression.
Part B: Change in Lee cGVHD Symptom Scale | Up to 36 weeks
  Change in Lee cGVHD symptom scale will be assessed. It is a participant reported improvement in symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (8):
- South Korea (8):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No